CLINICAL TRIAL: NCT01313208
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Etanercept in Subjects With Moderately Active Rheumatoid Arthritis Despite DMARD Therapy
Brief Title: Moderate Rheumatoid Arthritis (RA) With Etanercept (Enbrel)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20070561
Record Dates: First submitted 2011-03-10; First posted 2011-03-11 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Rheumatoid Arthritis
Keywords: RA; Enbrel; DMARD; Joint Count; Rheumatoid Arthritis; Etanercept; disease modifying anti-rheumatic drug
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo subcutaneous injections once a week for 12 weeks and then open-label etanercept 50 mg subcutaneous injection once weekly for the next 12 weeks.
  All participants continued their disease modifying anti-rheumatic drug (DMARD) treatment throughout the 24-week study period.
  Interventions: Drug: etanercept; Drug: Placebo; Drug: DMARD Therapy
- Etanercept (Experimental): Participants received etanercept 50 mg subcutaneous injection once weekly for 12 weeks and then open-label etanercept 50 mg subcutaneous injection for the next 12 weeks.
  All participants continued their DMARD treatment throughout the 24-week study period.
  Interventions: Drug: etanercept; Drug: DMARD Therapy

INTERVENTIONS:
Drug: etanercept — Administered by subcutaneous injection once weekly.
  Other Names: Enbrel
Drug: Placebo — Placebo subcutaneous injection
  Arms: Placebo
Drug: DMARD Therapy — Standard-of-care DMARD therapy, including methotrexate, sulfasalazine, leflunomide, minocycline, and/or hydroxychloroquine

SUMMARY:
This study is designed to evaluate the effectiveness of adding etanercept to disease modifying anti-rheumatic drug (DMARD) therapy in patients with moderately active Rheumatoid Arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 and ≤80 years of age at time of screening
* Diagnosed with rheumatoid arthritis as determined by meeting 1987 American College of Rheumatology (ACR) classification criteria and has had rheumatoid arthritis for at least 6 months
* Moderate rheumatoid arthritis during screening, as defined by a disease activity score (28 joint) calculated using the C-reactive protein formula (DAS28-CRP) > 3.2 and ≤ 5.1
* Active rheumatoid arthritis defined as ≥ 3 swollen joints (out of 28 joints examined) and ≥ 3 tender/painful joints (out of 28 joints examined) at screening and baseline. (A full 66/68 count joint count will be performed at baseline, but only joints in the 28-count joint count will be considered for eligibility. The 28-joint count consists of the finger joints excluding the distal interphalangeal joints, the wrists, elbows, shoulders, and knees)
* Must be currently taking a DMARD such as methotrexate, sulfasalazine, leflunomide, minocycline, and/or hydroxychloroquine

Exclusion Criteria:

* Prosthetic joint infection within 5 years of screening or native joint infection within 1 year of screening
* Class IV rheumatoid arthritis according to ACR revised response criteria
* Any active infection (including chronic or localized infections) for which anti-infectives were indicated within 28 days prior to first investigational product dose
* Previously used more than one experimental biologic DMARD. Patient with prior use of no more than one experimental biologic is permitted if the subject received no more than 8 weeks of treatment. The use of the experimental biologic must not have occurred within 2 months of the first dose of investigational product
* Previously used more than one commercially available biologic DMARD. Subject with prior use of no more than one commercially available biologic is permitted if the patient received no more than 8 weeks of treatment and did not discontinue because of lack of effect. The use of the biologic must not have occurred within 2 months of the first dose of investigational product. Acceptable prior use of biologics include the following examples:
* No more than 4 injections of adalimumab
* No more than 8 (50 mg) injections of etanercept
* No more than 2 infusions of infliximab
* No more than 2 infusions of abatacept
* Additional inclusion (exclusion) criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2011-03; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (44):
- United States (37):
  - Research Site, Birmingham, Alabama
  - Research Site, Tuscaloosa, Alabama
  - Research Site, Peoria, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Encino, California
  - Research Site, Hemet, California
  - Research Site, Inglewood, California
  - Research Site, La Jolla, California
  - Research Site, Murrieta, California
  - Research Site, Santa Maria, California
  - Research Site, Tustin, California
  - Research Site, Upland, California
  - Research Site, Victorville, California
  - Research Site, Denver, Colorado
  - Research Site, Jacksonville, Florida
  - Research Site, Ocala, Florida
  - Research Site, Sarasota, Florida
  - Research Site, Sebring, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Meridian, Idaho
  - Research Site, Springfield, Illinois
  - Research Site, Lexington, Kentucky
  - Research Site, Frederick, Maryland
  - Research Site, Lansing, Michigan
  - Research Site, Saint Clair Shores, Michigan
  - Research Site, Bismarck, North Dakota
  - Research Site, Akron, Ohio
  - Research Site, Mayfield Village, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Erie, Pennsylvania
  - Research Site, Greer, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Chesapeake, Virginia
  - Research Site, Seattle, Washington
- Canada (7):
  - Research Site, Winnipeg, Manitoba
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Burlington, Ontario
  - Research Site, Laval, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Eustache, Quebec

REFERENCES:
- [Background] Hobbs K, Deodhar A, Wang B, Bitman B, Nussbaum J, Chung J, Collier DH. Randomized, double-blind, placebo-controlled study to evaluate the efficacy and safety of etanercept in patients with moderately active rheumatoid arthritis despite DMARD therapy. Springerplus. 2015 Mar 5;4:113. doi: 10.1186/s40064-015-0895-9. eCollection 2015. PMID 25793152
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled on 31 March 2011; Last patient enrolled 29 November 2012
Period: Double-blind Phase (Weeks 1 - 12)
Arm/Group | Placebo | Etanercept
Started | 104 | 106
Completed | 98 | 101
Not Completed | 6 | 5
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Adverse Event | 1 | 2
Not completed — Ineligibility determined | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Noncompliance | 1 | 0
Period: Open-label Phase (Weeks 13 - 24)
Arm/Group | Placebo | Etanercept
Started | 98 | 101
Completed | 92 | 98
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Noncompliance | 0 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Etanercept | Total
Number analyzed (Participants) | 104 | 106 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (12.8) | 56.5 (12.1) | 56.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 75 | 161
  Male | 18 | 31 | 49
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 2 | 5
  Black or African American | 8 | 9 | 17
  Mixed race | 1 | 0 | 1
  White | 90 | 91 | 181
  Other | 1 | 4 | 5
Duration of Rheumatoid Arthritis [Mean (Standard Deviation); unit: years] | 7.41 (8.11) | 8.26 (11.16) | 7.84 (9.76)
Baseline methotrexate use [Number; unit: participants]
  Yes | 93 | 94 | 187
  No | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving DAS28 Low Disease Activity at Week 12
Description: Low disease activity is defined by a disease activity score (28 joint) calculated using the C-reactive protein formula (DAS28-CRP) of less than 3.2. The DAS28 is a composite score to measure disease activity in patients with rheumatoid arthritis, derived from the following variables: • The number of swollen and tender joints assessed using the 28-joint count; • C-Reactive Protein (CRP) level • Patient's global assessment of disease activity measured on a likert scale from 0 (no activity at all) to 10 (worst activity).
  The DAS28 score ranges from zero up to approximately ten. DAS28 scores above 5.1 indicate high disease activity.
Time Frame: Week 12
Population: Primary analysis set (all randomized participants); last observation carried forward (LOCF) imputation was used.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants received placebo subcutaneous injections once a week for 12 weeks.
- Etanercept: Participants received etanercept 50 mg subcutaneous injection once weekly for 12 weeks.
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
percentage of participants | 21.2 | 33.0
Statistical Analysis 1: Comparison: Placebo vs Etanercept; Test type: Superiority or Other; p = 0.055, Mantel Haenszel; P-value from Mantel-Haenszel test stratified by participant's baseline methotrexate use (yes or no); Odds Ratio (OR) = 1.83, 95% CI 2-sided [0.99 to 3.41] — Etanercept/Placebo

2. Secondary Outcome: Percentage of Participants Achieving DAS28 Remission at Week 12
Description: Remission is defined by a DAS28 score less than 2.6. The DAS28 is a composite score to measure disease activity in patients with rheumatoid arthritis, derived from the following variables:
  * The number of swollen and tender joints assessed using the 28-joint count;
  * C-reactive protein (CRP)
  * Patient's global assessment of disease activity measured on a likert scale from 0 (no activity at all) to 10 (worst activity).
  The DAS28 score ranges from zero to ten. DAS28 above 5.1 indicates high disease activity.
Time Frame: Week 12
Population: Primary analysis set; LOCF was used
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
percentage of participants | 11.5 | 18.9

3. Secondary Outcome: Percentage of Participants Achieving DAS28 Low Disease Activity at All Other Timepoints
Description: Low disease activity is defined by a disease activity score (28 joint) calculated using the C-reactive protein formula (DAS28-CRP) of less than 3.2. The DAS28 is a composite score to measure disease activity in patients with rheumatoid arthritis, derived from the following variables:
  * The number of swollen and tender joints assessed using the 28-joint count;
  * C-Reactive Protein (CRP) level
  * Patient's global assessment of disease activity measured on a likert scale from 0 (no activity at all) to 10 (worst activity).
  The DAS28 score ranges from zero up to approximately ten. DAS28 scores above 5.1 indicate high disease activity.
Time Frame: Baseline and Weeks 2, 4, 8, 16, 20 and 24
Population: Primary analysis set; LOCF was used. "N" indicates the number of participants included in the analysis at each time point.
Measure: Number; unit: percentage of participants
Groups:
- Placebo: Participants received placebo subcutaneous injections once a week for 12 weeks and then etanercept 50 mg subcutaneous injection once weekly for the next 12 weeks.
- Etanercept: Participants received etanercept 50 mg subcutaneous injection once weekly for 12 weeks and then etanercept 50 mg once weekly for the next 12 weeks.
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
percentage of participants
  Baseline (N=104, 104) | 2.9 | 1.0
  Week 2 (N=99, 105) | 10.1 | 21.0
  Week 4 (N=104, 106) | 15.4 | 24.5
  Week 8 (N=104, 106) | 16.3 | 34.0
  Week 16 (N=104, 106) | 37.5 | 40.6
  Week 20 (N=104, 106) | 46.2 | 45.3
  Week 24 (N=104, 106) | 43.3 | 50.0

4. Secondary Outcome: Percentage of Participants Achieving DAS28 Remission at All Other Timepoints
Description: Remission is defined by a DAS28 score less than 2.6. The DAS28 is a composite score to measure disease activity in patients with rheumatoid arthritis, derived from the following variables:
  * The number of swollen and tender joints assessed using the 28-joint count;
  * C-reactive protein (CRP)
  * Patient's global assessment of disease activity measured on a likert scale from 0 (no activity at all) to 10 (worst activity).
  The DAS28 score ranges from zero to ten. A DAS28 above 5.1 indicates high disease activity.
Time Frame: Baseline and Weeks 2, 4, 8, 16, 20 and 24
Population: Primary analysis set; LOCF was used. "N" indicates the number of participants included in the analyses at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
percentage of participants
  Baseline (N=104, 104) | 1.0 | 0.0
  Week 2 (N=99, 105) | 5.1 | 8.6
  Week 4 (N=104, 106) | 6.7 | 11.3
  Week 8 (N=104, 106) | 5.8 | 25.5
  Week 16 (N=104, 106) | 22.1 | 25.5
  Week 20 (N=104, 106) | 29.8 | 26.4
  Week 24 (N=104, 106) | 32.7 | 31.1

5. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 20 Response at Each Timepoint
Description: A participant was a responder if the following 3 criteria for improvement from Baseline were met: • ≥ 20% improvement in tender joint count; • ≥ 20% improvement in swollen joint count; and • ≥ 20% improvement in at least 3 of the 5 following parameters: ◦ Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]); ◦ Patient's global assessment of disease activity (measured on a likert scale from 0 to 10); ◦ Physician's global assessment of disease activity (measured on a likert scale from 0 to 10); ◦ Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]); ◦ C-Reactive Protein level.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: Primary analysis set; LOCF was used. "N" indicates the number of participants with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
percentage of participants
  Week 2 (N=101, 105) | 14.9 | 28.6
  Week 4 (N=104, 106) | 19.2 | 36.8
  Week 8 (N=104, 106) | 23.1 | 50.0
  Week 12 (N=104, 106) | 28.8 | 40.6
  Week 16 (N=104, 106) | 47.1 | 49.1
  Week 20 (N=104, 106) | 54.8 | 51.9
  Week 24 N=104, 106) | 46.2 | 50.0

6. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 50 Response at Each Timepoint
Description: A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 50% improvement in tender joint count;
  * ≥ 50% improvement in swollen joint count; and
  * ≥ 50% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a likert scale from 0 to 10);
    * Physician's global assessment of disease activity (measured on a likert scale from 0 to 10);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * C-reactive protein (CRP) level.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: Primary analysis set; LOCF was used. "N" indicates the number of participants with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
percentage of participants
  Week 2 (N=101, 106) | 3.0 | 5.7
  Week 4 (N=104, 106) | 4.8 | 13.2
  Week 8 (N=104, 106) | 4.8 | 19.8
  Week 12, (N=104, 106) | 12.5 | 20.8
  Week 16 (N=104, 106) | 22.1 | 30.2
  Week 20 (N=104, 106) | 28.8 | 29.2
  Week 24 (N=104, 106) | 28.8 | 33.0

7. Secondary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 70 Response at Each Timepoint
Description: A participant was a responder if the following 3 criteria for improvement from Baseline were met:
  * ≥ 70% improvement in tender joint count;
  * ≥ 70% improvement in swollen joint count; and
  * ≥ 70% improvement in at least 3 of the 5 following parameters:
    * Patient's assessment of pain (measured on a 100 mm visual analog scale [VAS]);
    * Patient's global assessment of disease activity (measured on a likert scale from 0 to 10);
    * Physician's global assessment of disease activity (measured on a likert scale from 0 to 10);
    * Patient's self-assessment of physical function (Health Assessment Questionnaire - Disability Index [HAQ-DI]);
    * C-reactive protein (CRP) level.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: Primary analysis set; LOCF was used. "N" indicates the number of participants with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
percentage of participants
  Week 2 (N=101, 106) | 0.0 | 1.9
  Week 4 (N=104, 106) | 0.0 | 1.9
  Week 8 (N=104, 106) | 0.0 | 5.7
  Week 12, (N=104, 106) | 1.0 | 5.7
  Week 16 (N=104, 106) | 9.6 | 8.5
  Week 20 (N=104, 106) | 10.6 | 17.0
  Week 24 (N=104, 106) | 12.5 | 16.0

8. Secondary Outcome: Percentage of Participants With RAPID3 Remission or Low Severity at Each Time Point
Description: The Multi-Dimensional Health Assessment Questionnaire (MDHAQ) is adapted from the standard HAQ and is used for the computation of the Routine Assessment of Patient Index Data 3 (RAPID3). The RAPID 3 includes the 3 Core Data Set measures of physical function, pain, and patient global estimate. The score for physical function ranges from 0 to 10 and is calculated by adding the ten activities of daily living, each scored from 0 to 3 by the patient (0="without any difficulty", 1="with some difficulty", 2="with much difficulty", and 3="unable to do") and dividing the total raw score by 3. Pain and global estimate of health are measured on a likert scale from 0 to 10, both scored 0 (best) to 10 (worst). The three 0-10 scores for physical function, pain, and global assesment of health are added together for a composite score of 0 to 30. The RAPID3 composite score includes 4 categories: High Severity > 12, Moderate Severity = 6.1 - 12, Low severity = 3.1 - 6, and Remission ≤ 3.
Time Frame: Baseline and Weeks 4, 12, and 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
percentage of participants
  Baseline (N=96, 99) | 9.4 | 9.1
  Week 4 (N=95, 99) | 21.1 | 30.3
  Week 12 (N=102, 103) | 21.6 | 39.8
  Week 24 (N=103, 103) | 41.7 | 46.6

9. Secondary Outcome: Percentage of Participants Achieving Count Remission at Each Time Point
Description: Count remission is achieved when a participant satisfies all of the following at any given time point: - 68 tender joint count ≤ 1, - 66 swollen joint count ≤ 1, - C-reactive protein (CRP) (in mg/dL) ≤1, and - patient global assessment of disease activity ≤ 1 (measured on a likert scale from 0 to 10 ranging from "no activity at all" to "worst activity imaginable").
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
percentage of participants
  Baseline (N=104, 106) | 0.0 | 0.0
  Week 2 (N=101, 106) | 1.0 | 0.0
  Week 4 (N=104, 106) | 0.0 | 2.8
  Week 8 (N=104, 106) | 0.0 | 2.8
  Week 12 (N=104, 106) | 1.9 | 4.7
  Week 16 (N=104, 106) | 3.8 | 5.7
  Week 20 (N=104, 106) | 5.8 | 10.4
  Week 24 (N=104, 106) | 7.7 | 10.4

10. Secondary Outcome: Percentage of Participants Achieving CDAI Remission at Each Time Point
Description: The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the:
  * 28 tender joint count (TJC),
  * 28 swollen joint count (SJC),
  * Patient's Global Assessment of Disease Activity measured on a likert scale from 0 to 10, where 0 = lowest disease activity and 10 = highest;
  * Physician's Global Assessment of Disease Activity measured on a Likert scale from 0 to 10, where 0 = lowest disease activity and 10 = highest.
  The CDAI score ranges from 0-76 where lower scores indicate less disease activity. CDAI remission is defined as a score ≤ 2.8.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
percentage of participants
  Baseline (N=101, 101) | 0.0 | 0.0
  Week 2 (N=99, 106) | 1.0 | 1.9
  Week 4 (N=104, 106) | 0.0 | 0.9
  Week 8 (N=104, 106) | 0.0 | 2.8
  Week 12 (N=104, 106) | 1.0 | 3.8
  Week 16 (N=104, 106) | 3.8 | 7.5
  Week 20 (N=104, 106) | 6.7 | 10.4
  Week 24 (N=104, 106) | 3.8 | 8.5

11. Secondary Outcome: Percentage of Participants Achieving CDAI Low Disease Activity at Each Time Point
Description: The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the:
  * 28 tender joint count (TJC),
  * 28 swollen joint count (SJC),
  * Patient's Global Assessment of Disease Activity measured on a Likert scale form 0 to 10, where 0 = lowest disease activity and 10 = highest;
  * Physician's Global Assessment of Disease Activity -measured on a Likert scale from 0 to 10, where 0 = lowest disease activity and 10 = highest. The CDAI score ranges from 0 to 76 where lower scores indicate less disease activity. CDAI low disease activity is defined as a score ≤ 10.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
percentage of participants
  Baseline (N=101, 101) | 0.0 | 0.0
  Week 2 (N=99, 106) | 9.1 | 12.3
  Week 4 (N=104, 106) | 16.3 | 18.9
  Week 8 (N=104, 106) | 15.4 | 29.2
  Week 12 (N=104, 106) | 21.2 | 25.5
  Week 16 (N=104, 106) | 32.7 | 35.8
  Week 20 (N=104, 106) | 42.3 | 38.7
  Week 24 (N=104, 106) | 41.3 | 46.2

12. Secondary Outcome: Clinical Disease Activity Index (CDAI) Score at Each Time Point
Description: The Clinical Disease Activity Index (CDAI) is a composite index that is calculated as the sum of the:
  * 28 tender joint count (TJC),
  * 28 swollen joint count (SJC),
  * Patient's Global Assessment of Disease Activity measured on a Likert scale from 0 to 10 where 0 = lowest disease activity and 10 = highest;
  * Physician's Global Assessment of Disease Activity (measured on a Likert scale from 0 to 10 where 0 = lowest disease activity and 10 = highest).
  The CDAI score ranges from 0 to 76 where lower scores indicate less disease activity.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Baseline (N=101, 101) | 30.18 (9.30) | 29.79 (9.08)
  Week 2 (N=99, 106) | 26.67 (12.89) | 24.32 (12.94)
  Week 4 (N=104, 106) | 24.81 (12.76) | 21.56 (12.82)
  Week 8 (N=104, 106) | 22.83 (12.25) | 20.22 (13.96)
  Week 12 (N=104, 106) | 22.79 (14.07) | 20.68 (14.90)
  Week 16 (N=104, 106) | 18.03 (12.34) | 18.28 (15.16)
  Week 20 (N=104, 106) | 15.13 (10.80) | 17.47 (14.90)
  Week 24 (N=104, 106) | 16.33 (11.85) | 16.86 (14.74)

13. Secondary Outcome: Percentage of Participants Achieving SDAI Remission at Each Time Point
Description: The simplified disease activity index (SDAI) is a composite measure that sums the total number of:
  * 28 tender joint counts,
  * 28 swollen joint counts,
  * Patient's Global Assessment of Disease Activity measured on a Likert scale from 0 to 10 where 0= lowest disease activity and 10 = highest;
  * Physician's Global Assessment of Disease Activity measured on a Likert scale from 0 to 10, where 0 = lowest disease activity and 10 = highest, and
  * C-reactive protein (CRP) in mg/dL.
  The SDAI score ranges from 0 to approximately 86 where lower scores indicate less disease activity. SDAI remission is defined as a score ≤ 3.3.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
percentage of participants
  Baseline (N=101, 101) | 0.0 | 0.0
  Week 2 (N=97, 105) | 1.0 | 1.0
  Week 4 (N=104, 106) | 1.0 | 0.9
  Week 8 (N=104, 106) | 0.0 | 5.7
  Week 12 (N=104, 106) | 1.9 | 5.7
  Week 16 (N=104, 106) | 4.8 | 8.5
  Week 20 (N=104, 106) | 8.7 | 11.3
  Week 24 (N=104, 106) | 6.7 | 10.4

14. Secondary Outcome: Percentage of Participants Achieving SDAI Low Disease Activity at Each Time Point
Description: The simplified disease activity index (SDAI) is a composite measure that sums the total number of: - 28 tender joint counts, - 28 swollen joint counts, - Patient's Global Assessment of Disease Activity measured on a Likert scale from 0 to 10 where 0 = lowest disease activity and 10 = highest; - Physician's Global Assessment of Disease Activity measured on a Likert scale from 0 to 10 where 0 = lowest disease activity and 10 = highest, and - C-reactive protein (CRP) in mg/dL. The SDAI score ranges from 0 to approximately 86 where lower scores indicate less disease activity. SDAI low disease activity is defined as a score ≤ 11.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
percentage of participants
  Baseline (N=101, 101) | 0.0 | 0.0
  Week 2 (N=97, 105) | 8.2 | 12.4
  Week 4 (N=104, 106) | 13.5 | 18.9
  Week 8 (N=104, 106) | 14.4 | 30.2
  Week 12 (N=104, 106) | 21.2 | 23.6
  Week 16 (N=104, 106) | 32.7 | 35.8
  Week 20 (N=104, 106) | 42.3 | 38.7
  Week 24 (N=104, 106) | 39.4 | 45.3

15. Secondary Outcome: Simplified Clinical Disease Activity Index (SDAI) Score at Each Time Point
Description: The simplified disease activity index (SDAI) is a composite measure that sums the total number of:
  * 28 tender joint counts,
  * 28 swollen joint counts,
  * Patient's Global Assessment of Disease Activity measured on a Likert scale from 0 to 10, where 0 = lowest disease activity and 10 = highest;
  * Physician's Global Assessment of Disease Activity measured on a Likert scale from 0 to 10, where 0 = lowest disease activity and 10 = highest, and
  * C-reactive protein (CRP) in mg/dL.
  The SDAI score ranges from 0 to approximately 86 where lower scores indicate less disease activity.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Baseline (N=101, 101) | 31.00 (9.49) | 30.56 (9.01)
  Week 2 (N=97, 105) | 27.83 (12.89) | 24.77 (12.96)
  Week 4 (N=104, 106) | 25.81 (12.89) | 22.00 (12.86)
  Week 8 (N=104, 106) | 23.64 (12.32) | 20.51 (14.08)
  Week 12 (N=104, 106) | 23.52 (14.02) | 21.09 (15.05)
  Week 16 (N=104, 106) | 18.55 (12.43) | 18.68 (15.25)
  Week 20 (N=104, 106) | 15.61 (10.77) | 17.87 (14.98)
  Week 24 (N=104, 106) | 16.93 (11.90) | 17.30 (14.85)

16. Secondary Outcome: Tender 28-Joint Count (TJC28) at Each Time Point
Description: Twenty-eight joints were assessed and classified as tender/not tender by pressure and joint manipulation on physical examination.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
tender joints
  Baseline (N=104, 106) | 11.1 (5.5) | 10.6 (5.1)
  Week 2 (N=101, 106) | 10.1 (6.7) | 9.6 (7.6)
  Week 4 (N=104, 106) | 9.4 (6.9) | 8.4 (6.9)
  Week 8 (N=104, 106) | 8.0 (6.2) | 7.7 (7.7)
  Week 12 (N=104, 106) | 8.8 (7.0) | 8.1 (8.0)
  Week 16 (N=104, 106) | 6.6 (6.3) | 6.9 (7.9)
  Week 20 (N=104, 106) | 5.1 (5.3) | 6.5 (7.9)
  Week 24 (N=104, 106) | 6.0 (6.4) | 6.5 (7.9)

17. Secondary Outcome: Swollen 28-Joint Count (SJC28) at Each Time Point
Description: Twenty-eight joints were assessed and classified as swollen/not swollen by pressure and joint manipulation on physical examination.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
swollen joints
  Baseline (N=104, 106) | 8.5 (4.4) | 8.4 (5.0)
  Week 2 (N=101, 106) | 6.9 (5.4) | 6.7 (4.5)
  Week 4 (N=104, 106) | 6.7 (5.3) | 5.4 (4.6)
  Week 8 (N=104, 106) | 6.2 (4.9) | 5.4 (4.9)
  Week 12 (N=104, 106) | 5.7 (5.4) | 5.5 (4.9)
  Week 16 (N=104, 106) | 5.0 (4.5) | 5.2 (5.4)
  Week 20 (N=104, 106) | 4.4 (4.7) | 4.8 (4.9)
  Week 24 (N=104, 106) | 4.6 (4.7) | 4.6 (5.2)

18. Secondary Outcome: Patient Global Assessment of Joint Pain at Each Time Point
Description: The severity of the participant's joint pain was assessed using a visual analog scale (VAS). The participant was asked to draw a mark through a 100 mm horizontal line to indicate how much pain they were experiencing "today", from '0' (no pain at all) on the left end of the line to 100 (worst pain imaginable) on the right end of the line.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Baseline (N=104, 106) | 43.74 (23.05) | 47.13 (23.22)
  Week 2 (N=101, 106) | 40.98 (23.58) | 33.41 (22.77)
  Week 4 (N=104, 106) | 38.65 (23.42) | 35.75 (24.92)
  Week 8 (N=104, 106) | 38.16 (23.64) | 31.18 (25.44)
  Week 12 (N=104, 106) | 38.38 (24.52) | 31.54 (26.46)
  Week 16 (N=104, 106) | 25.80 (20.52) | 28.97 (24.37)
  Week 20 (N=104, 106) | 23.98 (20.36) | 27.74 (25.83)
  Week 24 (N=104, 106) | 25.43 (22.12) | 28.09 (26.26)

19. Secondary Outcome: Patient's Global Assessment of Disease Activity at Each Time Point
Description: The participant's global assessment of their arthritis disease activity was assessed by the participant circling a number from 0 to 10 on a horizontal Likert scale ranging from "No Activity at All" (score = 0) to "Worst Activity Imaginable" (score = 10).
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Baseline (N=104, 106) | 5.0 (2.2) | 5.3 (2.1)
  Week 2 (N=101, 106) | 4.7 (2.3) | 4.0 (2.1)
  Week 4 (N=104, 106) | 4.5 (2.2) | 4.1 (2.3)
  Week 8 (N=104, 106) | 4.6 (2.3) | 3.7 (2.4)
  Week 12 (N=104, 106) | 4.3 (2.4) | 3.7 (2.5)
  Week 16 (N=104, 106) | 3.3 (2.2) | 3.3 (2.3)
  Week 20 (N=104, 106) | 2.9 (2.2) | 3.2 (2.6)
  Week 24 (N=104, 106) | 3.1 (2.2) | 3.1 (2.6)

20. Secondary Outcome: Physician Global Assessment of Disease Activity at Each Time Point
Description: The global assessment of the participant's arthritis was assessed by the physician circling a number from 0 to 10 on a horizontal Likert scale ranging from "No Activity at All" (score = 0) to "Worst Activity Imaginable" (score = 10).
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Baseline (N=101, 102) | 5.3 (1.7) | 5.4 (1.6)
  Week 2 (N=99, 106) | 4.6 (1.9) | 4.0 (1.8)
  Week 4 (N=104, 106) | 4.2 (1.9) | 3.7 (1.9)
  Week 8 (N=104, 106) | 4.0 (2.0) | 3.4 (2.1)
  Week 12 (N=104, 106) | 4.0 (2.1) | 3.3 (2.1)
  Week 16 (N=104, 106) | 3.1 (2.0) | 2.9 (2.0)
  Week 20 (N=104, 106) | 2.7 (1.7) | 2.9 (2.1)
  Week 24 (N=104, 106) | 2.7 (1.8) | 2.7 (1.9)

21. Secondary Outcome: Change From Baseline in the Disability Index of the Health Assessment Questionnaire (HAQ-DI) at Each Time Point
Description: The HAQ-DI asks about the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores). Responses in each functional area are scored from 0 indicating no difficulty to 3 indicating inability to perform a task in that area. The overall score is the average of each of the 8 category scores and ranges from 0 to 3, where zero represents no disability and three very severe, high-dependency disability.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: Primary analysis set; "N" indicates the number of participants included in the analyses at each time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Week 2 (N=98, 104) | -0.093 (0.385) | -0.266 (0.429)
  Week 4 (N=103, 105) | -0.164 (0.383) | -0.315 (0.528)
  Week 8 (N=99, 104) | -0.208 (0.420) | -0.370 (0.466)
  Week 12 (N=101, 101) | -0.203 (0.434) | -0.388 (0.543)
  Week 16 (N=98, 101) | -0.347 (0.476) | -0.403 (0.531)
  Week 20 (N=95, 97) | -0.412 (0.504) | -0.423 (0.578)
  Week 24 (N=91, 98) | -0.445 (0.522) | -0.475 (0.576)

22. Secondary Outcome: C-reactive Protein Levels at Each Time Point
Description: C-Reactive Protein (CRP) was measured from blood samples by a central laboratory as a marker for inflammation.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
mg/L
  Baseline (N=104, 106) | 9.44 (16.29) | 7.56 (11.77)
  Week 2 (N=100, 105) | 8.68 (11.49) | 3.97 (6.43)
  Week 4 (N=104, 106) | 9.75 (15.79) | 4.60 (8.27)
  Week 8 (N=104, 106) | 8.03 (10.26) | 3.94 (5.37)
  Week 12 (N=104, 106) | 8.33 (10.62) | 4.09 (6.11)
  Week 16 (N=104, 106) | 5.17 (7.58) | 3.76 (5.14)
  Week 20 (N=104, 106) | 4.75 (6.28) | 3.75 (4.55)
  Week 24 (N=104, 106) | 5.75 (13.10) | 4.40 (5.69)

23. Secondary Outcome: Short Form 36 Health Survey (SF-36) Physical Functioning Domain Score at Each Time Point
Description: The SF-36 measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). The individual domain scores are calculated and transformed to range from 0 to 100, with higher scores indicating a better level of functioning. The physical functioning subscale assesses limitations in physical activities because of health problems. Least Squares means are from a mixed-effect model for repeated measurements (MMRM).
Time Frame: Baseline and Weeks 4, 12 and 24
Population: Primary analysis set; Mixed-Effect Model Repeated Measures (MMRM) analysis to account for post-baseline missing data with Likelihood-based approach was used. "N" indicates the number of participants included in the analyses at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Baseline (N=100, 105) | 45.16 (2.75) | 45.71 (2.71)
  Week 4 (N=101, 102) | 47.54 (2.74) | 51.86 (2.72)
  Week 12 (N=99, 99) | 53.02 (2.75) | 52.06 (2.74)
  Week 24 (N=88, 97) | 60.38 (2.81) | 55.63 (2.75)

24. Secondary Outcome: Short Form 36 Health Survey (SF-36) Vitality Domain Score at Each Time Point
Description: The SF-36 measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). The individual domain scores are calculated and transformed to range from 0 to 100, with higher scores indicating a better level of functioning. The vitality sub-score assesses energy and fatigue. Least Squares means are from a mixed-effect model for repeated measurements (MMRM).
Time Frame: Baseline and Weeks 4, 12 and 24
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Baseline (N=101, 105) | 42.65 (2.14) | 41.11 (2.11)
  Week 4 (N=103, 105) | 46.45 (2.14) | 49.27 (2.12)
  Week 12 (N=100, 100) | 47.55 (2.15) | 48.90 (2.14)
  Week 24 (N=90, 98) | 53.03 (2.20) | 54.08 (2.15)

25. Secondary Outcome: Short Form 36 Health Survey (SF-36) Role-Physical Domain Score at Each Time Point
Description: The SF-36 measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). The individual domain scores are calculated and transformed to range from 0 to 100, with higher scores indicating a better level of functioning. The role-physical subscale assesses limitations in usual role activities because of physical health problems. Least squares means are from a mixed-effect model for repeated measurements (MMRM).
Time Frame: Baseline and Weeks 4, 12 and 24
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Baseline (N=104, 103) | 49.34 (2.74) | 51.69 (2.73)
  Week 4 (N=102, 105) | 56.09 (2.76) | 58.09 (2.72)
  Week 12 (N=100, 101) | 57.74 (2.77) | 57.83 (2.75)
  Week 24 (N=89, 97) | 65.87 (2.83) | 59.54 (2.77)

26. Secondary Outcome: Short Form 36 Health Survey (SF-36) Bodily Pain Domain Score at Each Time Point
Description: The SF-36 measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). The individual domain scores are calculated and transformed to range from 0 to 100, with higher scores indicating a better level of functioning (less pain). Least squares means are from a mixed-effect model for repeated measurements (MMRM).
Time Frame: Baseline and Weeks 4, 12 and 24
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Baseline (N=104, 106) | 41.98 (1.98) | 38.39 (1.96)
  Week 4 (N=103, 105) | 47.77 (1.99) | 52.17 (1.97)
  Week 12 (N=101, 101) | 51.15 (2.00) | 52.79 (1.99)
  Week 24 (N=88, 98) | 61.66 (2.08) | 59.42 (2.01)

27. Secondary Outcome: Short Form 36 Health Survey (SF-36) General Health Perceptions Domain Score at Each Time Point
Description: The SF-36 measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). The individual domain scores are calculated and transformed to range from 0 to 100, with higher scores indicating a better quality of life. Least squares means are from a mixed-effect model for repeated measurements (MMRM).
Time Frame: Baseline and Weeks 4, 12 and 24
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Baseline (N=104, 106) | 49.13 (2.03) | 51.77 (2.01)
  Week 4 (N=103, 104) | 52.52 (2.03) | 56.31 (2.02)
  Week 12 (N=100, 101) | 52.21 (2.04) | 54.77 (2.03)
  Week 24 (N=89, 98) | 55.94 (2.09) | 57.44 (2.04)

28. Secondary Outcome: Short Form 36 Health Survey (SF-36) Social Functioning Domain Score at Each Time Point
Description: The SF-36 measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). The individual domain scores are calculated and transformed to range from 0 to 100, with higher scores indicating a better level of functioning. The social functioning subscale assesses limitations in social activities because of physical or emotional problems. Least Squares means are from a mixed-effect model for repeated measurements (MMRM).
Time Frame: Baseline and Weeks 4, 12 and 24
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Baseline (N=104, 106) | 65.14 (2.61) | 63.21 (2.58)
  Week 4 (N=103, 105) | 69.04 (2.61) | 72.03 (2.59)
  Week 12 (N=101, 101) | 69.68 (12.62) | 69.32 (2.61)
  Week 24 (N=88, 98) | 78.59 (2.70) | 75.19 (2.63)

29. Secondary Outcome: Short Form 36 Health Survey (SF-36) Role-Emotional Domain Score at Each Time Point
Description: The SF-36 measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). The individual domain scores are calculated and transformed to range from 0 to 100, with higher scores indicating a better quality of life. The role-emotional subscale assesses limitations in usual role activities because of emotional problems. Least squares means are from a mixed-effect model for repeated measurements (MMRM).
Time Frame: Baseline and Weeks 4, 12 and 24
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Baseline (N=104, 104) | 69.23 (2.75) | 66.36 (2.74)
  Week 4 (N=102, 105) | 71.92 (2.77) | 72.56 (2.73)
  Week 12 (N=100, 100) | 75.86 (2.78) | 71.87 (2.77)
  Week 24 (N=89, 98) | 80.12 (2.86) | 76.30 (2.78)

30. Secondary Outcome: Short Form 36 Health Survey (SF-36) Mental Health Domain Score at Each Time Point
Description: The SF-36 measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). The individual domain scores are calculated and transformed to range from 0 to 100, with higher scores indicating a better quality of life. The mental health sub-score assesses general mental health (psychological distress and well-being). Least squares means are from a mixed-effect model for repeated measurements (MMRM).
Time Frame: Baseline and Weeks 4, 12 and 24
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Baseline (N=104, 104) | 70.14 (1.90) | 66.56 (1.88)
  Week 4 (N=103, 102) | 69.74 (1.90) | 72.01 (1.90)
  Week 12 (N=100, 100) | 72.05 (1.92) | 72.56 (1.90)
  Week 24 (N=89, 97) | 75.71 (1.96) | 74.20 (1.92)

31. Secondary Outcome: Work Productivity and Activity Impairment Questionnaire (WPAI): Percent Work Time Missed (Absenteeism) at Each Time Point
Description: This self-administered questionnaire is designed to address impairment to the work productivity and activity of participants due to rheumatoid arthritis in the past 7 days. Percent of work time missed is derived from the number of hours of work missed due to rheumatoid arthritis symptoms as a percentage of total hours that should have been worked. A higher percentage indicates more hours missed. Least squares means are from a mixed-effect model for repeated measurements (MMRM).
Time Frame: Baseline and Weeks 4, 12 and 24
Population: Primary analysis set; Mixed-Effect Model Repeated Measures (MMRM) analysis to account for post-baseline missing data with Likelihood-based approach was used. "N" indicates the number of participants employed and included in the analyses at each time point.
Measure: Least Squares Mean (Standard Error); unit: percent work time missed
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
percent work time missed
  Baseline (N=46, 46) | 3.54 (2.04) | 5.88 (2.03)
  Week 4 (N=46, 42) | 4.18 (2.03) | 4.50 (2.12)
  Week 12 (N=45, 40) | 8.07 (2.06) | 4.46 (2.16)
  Week 24 (N=38, 43) | 5.22 (2.21) | 3.77 (2.09)

32. Secondary Outcome: Work Productivity and Activity Impairment Questionnaire (WPAI): Percent Impairment While Working (Presenteeism) at Each Time Point
Description: This self-administered questionnaire is designed to address impairment to the work productivity and activity of participants due to rheumatoid arthritis in the past 7 days. Percent impairment while working was derived from the participant's assessment of the degree to which rheumatoid arthritis affected their productivity while working. A higher percentage indicates greater impairment and less productivity. Least squares means are from a mixed-effect model for repeated measurements (MMRM).
Time Frame: Baseline and Weeks 4, 12 and 24
Population: as for outcome 31
Measure: Least Squares Mean (Standard Error); unit: percent impairment while working
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
percent impairment while working
  Baseline (N=45, 45) | 34.39 (3.39) | 36.86 (3.39)
  Week 4 (N=44, 43) | 31.91 (3.41) | 25.04 (3.44)
  Week 12 (N=39, 40) | 25.49 (3.52) | 24.61 (3.50)
  Week 24 (N=37, 40) | 21.46 (3.57) | 21.10 (3.49)

33. Secondary Outcome: Work Productivity and Activity Impairment Questionnaire (WPAI): Percent Activity Impairment at Each Time Point
Description: This self-administered questionnaire is designed to address impairment to the work productivity and activity of participants due to rheumatoid arthritis. Percent activity impairment is derived from the patient's assessment of the degree to which rheumatoid arthritis affected their regular daily activities. A higher percentage indicates greater impairment and less productivity. Least squares means are from a mixed-effect model for repeated measurements (MMRM).
Time Frame: Baseline and Weeks 4, 12 and 24
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: percent activity impairment
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
percent activity impairment
  Baseline (N=103, 106) | 49.29 (2.56) | 50.38 (2.53)
  Week 4 (N=102, 104) | 41.22 (2.57) | 38.67 (2.55)
  Week 12 (N=99, 99) | 39.16 (2.59) | 35.98 (2.58)
  Week 24 (N=88, 96) | 29.91 (2.68) | 30.57 (2.61)

34. Secondary Outcome: Work Productivity and Activity Impairment Questionnaire (WPAI): Percent Overall Work Impairment at Each Time Point
Description: This self-administered questionnaire is designed to address impairment to the work productivity and activity of participants due to rheumatoid arthritis in the past 7 days. Percent overall work impairment takes into account both hours missed due to rheumatoid arthritis symptoms and the participant's assessment of the degree to which rheumatoid arthritis affected their productivity while working. A higher percentage indicates greater impairment and less productivity. Least squares means are from a mixed-effect model for repeated measurements (MMRM).
Time Frame: Baseline and Weeks 4, 12 and 24
Population: as for outcome 31
Measure: Least Squares Mean (Standard Error); unit: percent overall work impairment
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
percent overall work impairment
  Baseline (N=45, 46) | 34.79 (3.80) | 36.71 (3.76)
  Week 4 (N=46, 42) | 33.14 (3.77) | 26.14 (3.87)
  Week 12 (N=45, 40) | 27.23 (3.80) | 26.22 (3.92)
  Week 24 (N=38, 42) | 23.93 (3.98) | 22.58 (3.86)

35. Secondary Outcome: Participant Assessment of Fatigue at Each Time Point
Description: The participant's assessment of fatigue was collected using a single-item 100 mm visual analogue scale. The participant was asked to draw a vertical line through a horizontal line to indicate the degree of fatigue they experienced because of their condition over the past week. The horizontal line is 100 mm in length with '0' and 'no fatigue' on the left end of the line and '100' and 'extreme fatigue' on the right end of the line. Least squares means are from a mixed-effect model for repeated measurements (MMRM).
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Baseline (N=103, 105) | 49.38 (2.63) | 50.05 (2.61)
  Week 2 (N=99, 104) | 50.31 (2.66) | 38.68 (2.61)
  Week 4 (N=103, 105) | 46.48 (2.63) | 40.04 (2.61)
  Week 8 (N=99, 104) | 44.09 (2.66) | 39.32 (2.62)
  Week 12 (N=100, 100) | 45.51 (2.66) | 41.43 (2.64)
  Week 16 (N=98, 101) | 38.73 (2.67) | 35.15 (2.64)
  Week 20 (N=95, 97) | 29.82 (2.69) | 35.20 (2.66)
  Week 24 (N=90, 98) | 34.35 (2.72) | 33.87 (2.65)

36. Secondary Outcome: Medical Outcomes Study (MOS) Sleep Disturbance Scale at Each Time Point
Description: The MOS-Sleep comprises 12 items and measures key sleep structures across 6 domains. These domains are Sleep Disturbance (4 items), Sleep Adequacy (2 items), Sleep Quantity (1 item), Daytime Somnolence (3 items), Snoring (1 item), and Shortness of Breath (1 item). Sleep Disturbance measures the ability to fall asleep and to maintain restful sleep. In MOS Sleep norm-based scoring, all scales are scored on the same metric, where 50 is the mean for the general U.S. population and 10 is the standard deviation. Higher scores indicate more severe sleep problems. Least Squares means are from a mixed-effect model for repeated measurements (MMRM).
Time Frame: Baseline and Weeks 4, 12 and 24
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Baseline (N=102, 104) | 45.02 (1.00) | 44.95 (1.00)
  Week 4 (N=103, 104) | 46.42 (1.00) | 46.38 (1.00)
  Week 12 (N=98, 100) | 46.10 (1.01) | 46.91 (1.00)
  Week 24 (N=86, 96) | 48.23 (1.04) | 47.38 (1.01)

37. Secondary Outcome: Medical Outcomes Study (MOS) Sleep Shortness of Breath or Headache Scale at Each Time Point
Description: The MOS-Sleep comprises 12 items and measures key sleep structures across 6 domains. These domains are Sleep Disturbance (4 items), Sleep Adequacy (2 items), Sleep Quantity (1 item), Daytime Somnolence (3 items), Snoring (1 item), and Awakening short of breath or with a headache, (1 item). In MOS Sleep norm-based scoring, all scales are scored on the same metric, where 50 is the mean for the general U.S. population and 10 is the standard deviation. Higher scores indicate more severe sleep problems. Least Squares means are from a mixed-effect model for repeated measurements (MMRM).
Time Frame: Baseline and Weeks 4, 12 and 24
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Baseline (N=104, 106) | 51.63 (0.95) | 49.25 (0.94)
  Week 4 (N=103, 104) | 51.38 (0.95) | 50.20 (0.95)
  Week 12 (N=99, 98) | 50.34 (0.97) | 49.77 (0.97)
  Week 24 (N=89, 97) | 51.21 (1.00) | 50.31 (0.97)

38. Secondary Outcome: Medical Outcomes Study (MOS) Sleep Snoring Scale at Each Time Point
Description: The MOS-Sleep comprises 12 items and measures key sleep structures across 6 domains. These domains are Sleep Disturbance (4 items), Sleep Adequacy (2 items), Sleep Quantity (1 item), Daytime Somnolence (3 items), Snoring (1 item), and Shortness of Breath (1 item). In MOS Sleep norm-based scoring, all scales are scored on the same metric, where 50 is the mean for the general U.S. population and 10 is the standard deviation. Higher scores indicate more severe sleep problems. Least Squares means are from a mixed-effect model for repeated measurements (MMRM).
Time Frame: Baseline and Weeks 4, 12 and 24
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Baseline (N=101, 103) | 47.78 (0.95) | 47.13 (0.94)
  Week 4 (N=102, 102) | 49.14 (0.94) | 47.91 (0.94)
  Week 12 (N=99, 97) | 49.47 (0.95) | 49.04 (0.95)
  Week 24 (N=86, 93) | 49.95 (0.98) | 48.25 (0.96)

39. Secondary Outcome: Medical Outcomes Study (MOS) Sleep Adequacy Scale at Each Time Point
Description: The MOS-Sleep comprises 12 items and measures key sleep structures across 6 domains. These domains are Sleep Disturbance (4 items), Sleep Adequacy (2 items), Sleep Quantity (1 item), Daytime Somnolence (3 items), Snoring (1 item), and Awakening short of breath or with a headache, (1 item). Sleep Adequacy measures sleep sufficiency in terms of whether the participant sleeps enough to provide restoration of wakefulness. In MOS Sleep norm-based scoring, all scales are scored on the same metric, where 50 is the mean for the general U.S. population and 10 is the standard deviation. For sleep adequacy a higher score indicates better sleep quality. Least Squares means are from a mixed-effect model for repeated measurements (MMRM).
Time Frame: Baseline and Weeks 4, 12 and 24
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Baseline (N=102, 105) | 47.12 (0.98) | 46.72 (0.97)
  Week 4 (N=103, 104) | 47.63 (0.98) | 47.42 (0.97)
  Week 12 (N=99, 99) | 46.86 (0.99) | 47.73 (0.98)
  Week 24 (N=87, 97) | 48.73 (1.02) | 48.66 (0.99)

40. Secondary Outcome: Medical Outcomes Study (MOS) Sleep Daytime Somnolence Scale at Each Time Point
Description: The MOS-Sleep comprises 12 items and measures key sleep structures across 6 domains. These domains are Sleep Disturbance (4 items), Sleep Adequacy (2 items), Sleep Quantity (1 item), Daytime Somnolence (3 items), Snoring (1 item), and Awakening short of breath or with a headache, (1 item). Daytime somnolence measures drowsiness or sleepiness during the day. In MOS Sleep norm-based scoring, all scales are scored on the same metric, where 50 is the mean for the general U.S. population and 10 is the standard deviation. Higher scores indicate more severe sleep problems. Least Squares means are from a mixed-effect model for repeated measurements (MMRM).
Time Frame: Baseline and Weeks 4, 12 and 24
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Baseline (N=103, 106) | 46.82 (1.01) | 46.27 (1.00)
  Week 4 (N=103, 104) | 46.62 (1.01) | 48.72 (1.01)
  Week 12 (N=99, 99) | 47.80 (1.02) | 48.05 (1.02)
  Week 24 (N=87, 97) | 48.31 (1.05) | 48.80 (1.02)

41. Secondary Outcome: Medical Outcomes Study (MOS) Sleep Problems Index I at Each Time Point
Description: The MOS-Sleep comprises 12 items and measures key sleep structures across 6 domains. These domains are Sleep Disturbance (4 items), Sleep Adequacy (2 items), Sleep Quantity (1 item), Daytime Somnolence (3 items), Snoring (1 item), and Awakening short of breath or with a headache, (1 item). The scale also produces two indices. The Sleep Problems Index-I is drawn from 6 items in the four domains including Sleep Disturbance (2 items), Sleep Adequacy (2 items), Shortness of Breath (1 item), and Daytime Somnolence (1 item). In MOS Sleep norm-based scoring, all scales are scored on the same metric, where 50 is the mean for the general U.S. population and 10 is the standard deviation. Higher scores indicate more severe sleep problems. Least Squares means are from a mixed-effect model for repeated measurements (MMRM).
Time Frame: Baseline and Weeks 4, 12 and 24
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Baseline (N=102, 105) | 46.16 (0.92) | 45.53 (0.91)
  Week 4 (N=103, 104) | 46.91 (0.92) | 46.63 (0.91)
  Week 12 (N=99, 97) | 46.82 (0.92) | 47.17 (0.92)
  Week 24 (N=87, 97) | 48.39 (0.95) | 47.80 (0.92)

42. Secondary Outcome: Medical Outcomes Study (MOS) Sleep Problems Index II at Each Time Point
Description: The MOS-Sleep comprises 12 items and measures key sleep structures across 6 domains. These domains are Sleep Disturbance (4 items), Sleep Adequacy (2 items), Sleep Quantity (1 item), Daytime Somnolence (3 items), Snoring (1 item), and Awakening short of breath or with a headache, (1 item). The scale also produces two indices. Index-II uses 9 items from four domains including Sleep Disturbance (4 items), Sleep Adequacy (2 items), Shortness of Breath (1 item), and Daytime Somnolence (2 items). In MOS Sleep norm-based scoring, all scales are scored on the same metric, where 50 is the mean for the general U.S. population and 10 is the standard deviation. Higher scores indicate more severe sleep problems. Least Squares means are from a mixed-effect model for repeated measurements (MMRM).
Time Frame: Baseline and Weeks 4, 12 and 24
Population: as for outcome 23
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Etanercept
Number analyzed (Participants) | 104 | 106
scores on a scale
  Baseline (N=101, 104) | 45.69 (0.93) | 45.16 (0.92)
  Week 4 (N=103, 104) | 46.63 (0.93) | 48.84 (0.92)
  Week 12 (N=98, 97) | 46.51 (0.94) | 47.06 (0.94)
  Week 24 (N=86, 96) | 48.55 (0.96) | 47.88 (0.94)

ADVERSE EVENTS:
Time Frame: 28 weeks
Description: The table of Other Adverse Events summarizes non-serious occurrences of adverse events that exceeded a 5% frequency threshold in either treatment group.
Groups:
- Placebo-Etanercept: Participants received placebo subcutaneous injections once a week for 12 weeks and then open-label etanercept 50 mg subcutaneous injection once weekly for the next 12 weeks. All participants continued their disease modifying anti-rheumatic drug (DMARD) treatment throughout the 24-week study period.
- Etanercept-Etanercept: Participants received etanercept 50 mg subcutaneous injection once weekly for 12 weeks and then open-label etanercept 50 mg subcutaneous injection for the next 12 weeks. All participants continued their DMARD treatment throughout the 24-week study period.
Arm/Group | Placebo-Etanercept | Etanercept-Etanercept
Serious Adverse Events (participants affected / at risk) | 3/104 | 4/106
Other Adverse Events (participants affected / at risk) | 61/104 | 62/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Etanercept (N=104) | Etanercept-Etanercept (N=106)
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo-Etanercept (N=104) | Etanercept-Etanercept (N=106)
Nausea (Gastrointestinal disorders) | 6 | 5
Fatigue (General disorders) | 4 | 6
Injection site erythema (General disorders) | 11 | 13
Injection site pain (General disorders) | 6 | 5
Injection site pruritus (General disorders) | 8 | 7
Injection site rash (General disorders) | 6 | 9
Bronchitis (Infections and infestations) | 4 | 7
Nasopharyngitis (Infections and infestations) | 12 | 6
Sinusitis (Infections and infestations) | 7 | 8
Upper respiratory tract infection (Infections and infestations) | 13 | 8
Urinary tract infection (Infections and infestations) | 4 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 6
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 12 | 12
Headache (Nervous system disorders) | 16 | 9
Rash (Skin and subcutaneous tissue disorders) | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.